CLINICAL TRIAL: NCT05688722
Title: Head Elevation During Pre-oxygenation Can Delay Desaturation Time in Indonesian Patients
Brief Title: Head Elevation During Pre-oxygenation Can Delay Desaturation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ratna Farida Soenarto, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes913
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Surgery; Desaturation of Blood; Apnea
Keywords: preoxygenation; head elevation; desaturation; apnea
MeSH Terms: conditions — Apnea | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: Patients were divided into 4 groups by random sampling each with different intervention
Who Masked: Participant
Masking Description: The care provider and investigator were not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Patient positioned in supine conventional position
  Interventions: Procedure: Supine position
- 20 degree head elevation (Active Comparator): Patient positioned in 20 degree head elevation position
  Interventions: Procedure: 20 degree head elevation position
- 30 degree head elevation (Active Comparator): Patient positioned in 30 degree head elevation position
  Interventions: Procedure: 30 degree head elevation position
- 45 degree head elevation (Active Comparator): Patient positioned in 45 degree head elevation position
  Interventions: Procedure: 45 degree head elevation position

INTERVENTIONS:
Procedure: Supine position — Patients preoxygenated in supine position before endotracheal intubation
  Arms: Control
Procedure: 20 degree head elevation position — Patients preoxygenated in 20 degree head elevation position before endotracheal intubation
  Arms: 20 degree head elevation
Procedure: 30 degree head elevation position — Patients preoxygenated in 30 degree head elevation position before endotracheal intubation
  Arms: 30 degree head elevation
Procedure: 45 degree head elevation position — Patients preoxygenated in 45 degree head elevation position before endotracheal intubation
  Arms: 45 degree head elevation

SUMMARY:
This study is a randomized-controlled trial study comparing the association between several degree of head elevation and conventional position during pre-oxygenation to desaturation time in patients undergo endotracheal intubation with general anesthesia

DETAILED DESCRIPTION:
Preoxygenation anesthesia induction is an important part of airway management to reduce the risk of hypoxemia when the patient is apneic. The effectivity of preoxygenation is influenced by several things such as patient's head position. This study aimed to compare preoxygenation with head elevation 20°, 30° and 45° and conventional position to the time of desaturation before endotracheal intubation in patients undergoing general anesthesia. This was a randomized clinical trial of 56 patients, divided into four groups (conventional or 0° head elevation group, 20° head elevation group, 30° head elevation and 45° head elevation group). All subject was preoxygenated for 3 minutes with 100% oxygen. Induction of anesthesia was started with fentanyl, propofol, followed by rocuronium after the patient lost consciousness. Time was recorded from the start of induction until the oxygen saturation showed 93% or a time limit of 5 minutes. There was a significant difference in mean desaturation time among the four groups (p = 0.011). The most significant different was in 45o head elevation group (p < 0.05). . In patients undergoing general anesthesia, pre-oxygenation with head elevation 20°, 30° and 45° slows down the time for desaturation before endotracheal intubation compared to the conventional position. The 45° head elevation has the best result.

ELIGIBILITY:
Inclusion Criteria:

* undergo endotracheal intubation with general anesthesia for elective surgery
* aged 18-60 years old
* ASA physical status 1-2 preoperatively

Exclusion Criteria:

* Patients with difficult airway, cardiopulmonary disease, anemia, grade II obesity, pregnant, history of hypersensitivity to induction agents
* Patients did not give consent to follow the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Desaturation time | Right after induction until reach oxygen saturation 93% or 5 minutes time limit
  Time was recorded from the start of induction until the oxygen saturation showed 93% or a time limit of 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ratna F Soenarto, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia